CLINICAL TRIAL: NCT00385359
Title: A Pilot Efficacy Study of Inhaled Albuterol Delivered With Akita Breath Control and Pari Nebulization for the Treatment of Adults With Moderate Asthma
Brief Title: A Pilot Efficacy Study of Inhaled Albuterol Delivered With Akita Breath Control
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IA-01
Record Dates: First submitted 2006-10-06; First posted 2006-10-09 (Estimated); Last update posted 2006-10-09 (Estimated); Status verified 2006-10

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Albuterol

INTERVENTIONS:
Procedure: aerosol drug deposition strategies
Drug: Albuterol

SUMMARY:
Albuterol (salbutamol) is a widely used asthma medication but is associated with undesirable side effects such as shakiness and increased heart rate. Targeted delivery of albuterol to area of lungs where it has most effect would require a lower total dose to produce the same beneficial effects while reducing the side effects.

It is anticipated that only 1/13th to 1/25th of the standard nebulized dose of albuterol will be required to attain same bronchodilator response as a standard nebulizer treatment as determined by lung function measurement and that the reduced dose will significantly reduce side effects as determined by hand tremor and heart rate.

DETAILED DESCRIPTION:
Side effects of albuterol (salbutamol)are directly related to the dose delivered and absorbed into blood stream. By controlling aerosol delivery, dose delivered, site of deposition, amount of drug absorption can be determined and thus the magnitude of the side effects. Delivery and deposition of aerosols are determined by both aerosol characteristics (size and timing of delivery) and breathing characteristics (breath size, flow rate and breathholding). Data supports the theory that if a high dose of albuterol can be deposited in the larger airway generations and prevented from entering the pulmonary circulation from the lung periphery, that this will result in the largest magnitude of bronchodilator response with the lowest circulatory absorbance.

This is a pilot study in 10 adults with moderate asthma. there are no investigational drugs or devices. It is an investigation of a strategy to maximize response to an approved drug while minimizing side effects. The investigational strategies will deposit less than 25% of the standard nebulized dose in the airways. This will be accomplished by pairing a Pari eFlow nebulizer configured to deliver particle sizes of 3.5 to 6 microns, with an Akita delivery system programmed to deliver the drug as either a late or early bolus during inspiration. The Akita is programmed with a specific breathing pattern based on participant's lung function tests at screening.

Moderate asthmatics with bronchodilator response >20% improvement in FEV1 will be selected. Treatments will be administered on separate days 1-7 days apart. Following baseline measurements 1 of 5 randomized aerosol treatments will be administered. Efficacy (FEV1) and side effects (tremor and heart rate)will be monitored for 6 hours following drug administration.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-60 years
* Moderate asthma with baseline FEV1 40-75% predicted
* Previous use of albuterol (salbutamol)
* At least 20% improvement in FEV1 following 2.5 mg albuterol (salbutamol) delivered by nebulizer
* O2 saturation > 90%
* Non-smoker for > 6 months

Exclusion Criteria:

* Upper respiratory tract infection or asthma exacerbation within 14 days of screening
* Clinically significant abnormal chest radiograph
* History of cardiovascular disorder including coronary insufficiency, cardiac arrhythmias or hypertension
* Unable to tolerate bronchodilator withdrawal
* Known hypersensitivity to albuterol (salbutamol)
* Change in asthma treatment regimen in past 30 days

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10
Dates: Start 2006-10

PRIMARY OUTCOMES:
change in FEV1 expressed as a percent of predicted between baseline and 1 hour post drug administration.

SECONDARY OUTCOMES:
duration of effect based on FEV1 at 6 hours post treatment compared to standard treatment
change in hand tremor compared to standard treatment
change in heart rate compared to standard treatment

CONTACTS AND LOCATIONS:
Overall Officials: Victor Hoffstein, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital - Respiratory Research Lab, Toronto, Ontario, Canada